CLINICAL TRIAL: NCT05163080
Title: Prospective Randomized Placebo-Controlled Trial of SurVaxM Plus Adjuvant Temozolomide for Newly Diagnosed Glioblastoma (SURVIVE)
Brief Title: SurVaxM Plus Adjuvant Temozolomide for Newly Diagnosed Glioblastoma (SURVIVE)
Acronym: SURVIVE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MimiVax, LLC (Industry)
Collaborators: Translational Drug Development (Other); Merit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: I-813720
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Newly Diagnosed Glioblastoma

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, placebo-controlled, multi-center study of patients with newly diagnosed Glioblastoma (nGBM)to evaluate a peptide vaccine (SurVaxM) in emulsion with Montanide given together with locally administered sargramostim plus adjuvant oral temozolomide (Arm A) versus saline-Montanide emulsion with locally administered saline (instead of sargramostim) plus adjuvant oral temozolomide (Arm B)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Peptide Vaccine (SurVaxM) in emulsion with Montanide given together with locally administered Sargramostim plus adjuvant oral Temozolomide
  Interventions: Biological: SurVaxM
- Arm B (Placebo Comparator): Saline-Montanide emulsion with locally administered saline (instead of sargramostim) plus adjuvant oral temozolomide
  Interventions: Biological: SurVaxM

INTERVENTIONS:
Biological: SurVaxM — Consists of a synthetic peptide conjugate that stimulates immune responses capable of killing cancer cells that express the survivin molecule. Multiple copies of the multiplied peptide (SVN53-67/M57) are conjugated to Keyhole Limpet Hemocyanin (KLH) yielding a molecule designated as SVN53-67/M57-KLH. The SVN53-67/M57-KLH conjugate (SurVaxM)produces immune responses in mice and humans that are cross-reactive to the wild-type survivin molecule expressed by tumor cells. The survivin peptide in SurVaxM is a defined antigenic peptide comprised of 15 amino acids that encompass multiple epitopes capable of binding human MHC Class I and murine H2-Kb molecules. SurVaxM also contains a core antigenic epitope that has been modified by substitution of methionine for cysteine at amino acid position 57 (i.e., M57).

SUMMARY:
The main purpose of this study is to determine whether adding SurVaxM to standard-of-care temozolomide chemotherapy is better than temozolomide treatment alone for patients with newly diagnosed glioblastoma. This study is designed to compare the length of survival in patients with newly diagnosed glioblastoma who receive temozolomide plus SurVaxM to that of patients treated with standard-of-care temozolomide plus placebo. This study aims to discover what effects, both good and bad, this combination of drugs may have on you and to see if the study drug (SurVaxM) can create an immune response in your blood that is directed against your cancer cells. This study also aims to determine whether treatment with SurVaxM plus temozolomide improves the survival of glioblastoma patients like yourself compared to treatment with temozolomide alone.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled study. That means that some patients will receive an active drug (SurVaxM) and some will receive an inactive drug (placebo). Patients who agree to participate will be randomized (chance) to one of two groups. Patients that are randomized by chance to receive SurVaxM will be treated with standard-of-care temozolomide plus an injection under the skin of SurVaxM in Montanide (a milky white substance that helps SurVaxM to be recognized by the patient's immune system). Patients in this group will also receive a second separate injection of a drug called sargramostim that boosts the patient's immune system at the site of the first injection. These injections will be repeated at regular intervals according to a schedule.

Patients that are randomized to receive placebo will be treated with standard-of-care temozolomide plus an injection under the skin of saline (salt water) in Montanide (a milky white substance). Patients in this group will also receive a second separate injection of saline to simulate the injection of sargramostim that patient's in the SurVaxM group receive. These injections will be repeated at regular intervals according to a schedule.

The treatments in the two groups (SurVaxM and placebo groups) will be completely indistinguishable to patients and their treating doctors.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, participants must meet the following criteria:

1. Age ≥ 18 years of age.
2. Have a Karnofsky performance status ≥ 70 (i.e., the patient must be able to care for him/herself with occasional help from others; refer to Appendix A).

3 .Pathologically confirmed diagnosis of glioblastoma of the cerebrum.

4 .The result of tumor MGMT methylation study must be available.

5 .The result of tumor IDH-1 mutation test must be available.

6. Have the following clinical laboratory values obtained within 14 days prior to registration:

1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
2. Platelets ≥ 100 x 109/L
3. Hemoglobin (Hgb) ≥ 9.0 g/dL
4. Total bilirubin: ≤ 1.5 x ULN
5. ALT and AST ≤ 4.0 x ULN
6. Creatinine ≤ 1.8 mg/dL
7. Prothrombin time (PT) within 1.5x normal limits
8. Activated partial thromboplastin time (aPPT) within 1.5x control
9. International Normalized Ration (INR) less than or equal to 1.5x control

   7. Patient must have no active bleeding or pathological condition that carries a high risk of bleeding (e.g., coagulopathy)

   8. Available results from a contrast-enhanced, post-operative brain MRI that was completed within 72 hours after surgery documenting either:

a. gross total resection consisting of no gadolinium enhancement; or b. near-total resection consisting of either ≤ 1 cm3 nodular (i.e. volumetric) enhancement or ≤ 100 mm2 in cross sectional area (i.e. linear enhancement). Note: Patients who undergo either stereotactic biopsy or open biopsy for tissue diagnosis, or partial tumor resection, and who subsequently have a definitive surgical resection may still be eligible for inclusion, provided that randomization can occur within 16 weeks of the date of surgical resection. To be eligible, such patients must still meet postoperative imaging entry criteria as defined in item #8 above.

9. Patients must have completed initial radiation therapy with TMZ (chemoradiation) according to established Stupp protocol (Stupp, 2005) for the treatment of their glioblastoma (i.e., completed 6-week course of RT and completed ≥ 75% of a course of concurrent TMZ chemotherapy).

10. Patients must be randomized within 16 weeks of surgical resection of their newly diagnosed glioblastoma.

11. No evidence of progressive disease at the post-chemoradiation timepoint based on changes in: neurologic exam, corticosteroid use or radiographic progression (i.e., baseline MRI evaluation). (See Section 14.5 for suspected pseudo-progression.)

12. Participants of child-bearing potential (not surgically sterile or postmenopausal) must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and have a negative pregnancy test prior to starting study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

13. Dexamethasone dose less than or equal to 4 mg daily at time of study enrollment. Every reasonable effort should be made to reduce the dose of corticosteroids to the absolute minimum dose required to control neurologic symptoms prior to receiving SurVaxM.

14. Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

Participants with any of the following will be excluded from this study:

1. Recurrent or progressive glioblastoma.
2. Gliosarcoma, anaplastic astrocytoma, oligodendroglioma, ependymoma, low grade glioma or any histology other than glioblastoma.
3. Multicentric glioblastoma or glioblastoma involving the brainstem or cerebellum, or leptomeningeal or spinal extension present at diagnosis.
4. Residual contrast enhancement > 1 cm3 on post-operative scan obtained within 72 hours of surgery.
5. Absence of MRI obtained within 72 hours of craniotomy documenting

   ≤ 1 cm3 contrast-enhancing tumor.
6. Patients who elect to have Optune therapy (Tumor Treating Fields) are not eligible to participate in this trial.
7. Patient has had non-standard radiation therapy for glioblastoma (i.e., whole brain radiation therapy, gamma knife or LINAC stereotactic radiosurgery).
8. Prior or concurrent immunotherapy for brain tumor, including immune checkpoint inhibitors (pembrolizumab, nivolumab or ipilimumab) or other cancer vaccine therapy.
9. Prior or concurrent treatment with bevacizumab.
10. Patients with serious concurrent infection or medical illness, which in the treating physician's opinion would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety.
11. History of tuberculosis or other granulomatous disease.
12. Patient is pregnant or breast-feeding.
13. Patient has received any other chemotherapeutic agent or investigational drug in addition to standard of care radiation therapy with concomitant temozolomide (chemoradiation per Stupp protocol).
14. Patient with concurrent or prior malignancy is ineligible unless he or she has had curatively treated carcinoma-in-situ or basal cell carcinoma of the skin.
15. Patients who have had repeat craniotomy for tumor therapy after receiving RT and TMZ treatment (i.e., chemoradiation).
16. Patients who have had surgical implantation of carmustine (Gliadel) wafers are not eligible to participate in this study.
17. Known history of systemic autoimmune disorder.
18. Known human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS) related illness or other serious medical illness.
19. Patient has a contraindication to MRI scans or to gadolinium contrast agent.
20. Patient has a contraindication to temozolomide.
21. Patient is unwilling or unable to follow protocol requirements.
22. Patient has received any other investigational treatment for the glioblastoma.
23. Any condition which in the Investigator's opinion makes the candidate unsuitable to receive the study drug or protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-08-18 (Estimated); Study Completion 2024-08-18 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 36 Months
  To compare overall survival (OS) in patients with newly diagnosed glioblastoma between treatment arms A & B

SECONDARY OUTCOMES:
Grade 3 & Grade 4 Toxicities | 36 Months
  To tabulate the number and type of Grade 3 & Grade 4 toxicities, according to the NCI Common Toxicity Criteria for Adverse Events (NCI CTCAEs) Version 5
Progression Free Survival Comparison | 36 months
  To compare Progression Free Survival in patients with newly diagnosed glioblastoma between treatment arms A & B.
Overall Survival at Specified Time Points | 24 months
  To compare treatment-associated OS at pre-specified time points (OS-15, OS-18, and OS-24) between treatment arms A & B.
Progression-Free Survival at specific time points | 12 months
  To compare treatment associated PFS at pre-specified time points (PFS-3, PFS-6, PFS-12) between treatment arms A & B

OTHER OUTCOMES:
Predictive Value of perfusion-weighted imaging - pseudo-progression | 36 months
  To evaluate the predictive value of perfusion-weighted imaging in assessing pseudo-progression and post-vaccination enhancement in patents receiving SurVaxM
Objective Image Based Tumor Response Rate | 36 months
  To evaluate the objective image based tumor response rate (applicable only for patients with valuable disease at study entry as defined by RANO criteria)
Evaluate molecular predictors of response to SurVaxM | 36 months
  To evaluate the molecular predictors of response to SurVaxM, including MGMT methylation status, anti-surviving immunoglobin titers, surviving-specific CD8+ responses, tumor survivin expression levels and other molecular tumor tissue markers

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fenstermaker, MD, Principal Investigator — Chief Medical Officer; Michael Ciesielski, PhD, Study Director — Chief Executive Officer; Manmeet S Ahluwalia, MD, MBA, Principal Investigator — Study Principal Investigator
Locations (11):
- United States (11):
  - University of California, San Francisco, California
  - Miami Cancer Institute, Miami, Florida
  - Norton Cancer Center, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Atlantic Health, Summit, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - NYU Langone Health, New York, New York
  - Northwell, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Texas Oncology, Austin, Texas
  - Fred Hutchinson Cancer Center (FHCC), Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Result] Ciesielski MJ, Ahluwalia MS, Munich SA, Orton M, Barone T, Chanan-Khan A, Fenstermaker RA. Antitumor cytotoxic T-cell response induced by a survivin peptide mimic. Cancer Immunol Immunother. 2010 Aug;59(8):1211-21. doi: 10.1007/s00262-010-0845-x. Epub 2010 Apr 27. PMID 20422411
- [Result] Andersen MH, Pedersen LO, Becker JC, Straten PT. Identification of a cytotoxic T lymphocyte response to the apoptosis inhibitor protein survivin in cancer patients. Cancer Res. 2001 Feb 1;61(3):869-72. PMID 11221872
- [Result] Hadrup SR, Gehl J, Sorensen RB, Geertsen PF, Straten PT, Andersen MH. Persistence of survivin specific T cells for seven years in a melanoma patient during complete remission. Cancer Biol Ther. 2006 May;5(5):480-2. doi: 10.4161/cbt.5.5.2652. Epub 2006 May 5. PMID 16582593
- [Result] Baxevanis CN, Voutsas IF, Tsitsilonis OE, Gritzapis AD, Sotiriadou R, Papamichail M. Tumor-specific CD4+ T lymphocytes from cancer patients are required for optimal induction of cytotoxic T cells against the autologous tumor. J Immunol. 2000 Apr 1;164(7):3902-12. doi: 10.4049/jimmunol.164.7.3902. PMID 10725753
- [Result] Moeller M, Kershaw MH, Cameron R, Westwood JA, Trapani JA, Smyth MJ, Darcy PK. Sustained antigen-specific antitumor recall response mediated by gene-modified CD4+ T helper-1 and CD8+ T cells. Cancer Res. 2007 Dec 1;67(23):11428-37. doi: 10.1158/0008-5472.CAN-07-1141. PMID 18056471
- [Result] Yu J, Ren X, Cao S, Zhang W, Hao X. Th1 polarization and apoptosis-inducing activity of CD4+ T -cells in cytokine-induced killers might favor the antitumor cytotoxicity of cytokine-induced killers in vivo. Cancer Biother Radiopharm. 2006 Jun;21(3):276-84. doi: 10.1089/cbr.2006.21.276. PMID 16918305
- [Result] Surman DR, Dudley ME, Overwijk WW, Restifo NP. Cutting edge: CD4+ T cell control of CD8+ T cell reactivity to a model tumor antigen. J Immunol. 2000 Jan 15;164(2):562-5. doi: 10.4049/jimmunol.164.2.562. PMID 10623795
- [Result] Hung K, Hayashi R, Lafond-Walker A, Lowenstein C, Pardoll D, Levitsky H. The central role of CD4(+) T cells in the antitumor immune response. J Exp Med. 1998 Dec 21;188(12):2357-68. doi: 10.1084/jem.188.12.2357. PMID 9858522
- [Result] Pardoll DM. Inducing autoimmune disease to treat cancer. Proc Natl Acad Sci U S A. 1999 May 11;96(10):5340-2. doi: 10.1073/pnas.96.10.5340. No abstract available. PMID 10318881
- [Result] Fenstermaker RA, Figel SA, Qiu J, Barone TA, Dharma SS, Winograd EK, Galbo PM, Wiltsie LM, Ciesielski MJ. Survivin Monoclonal Antibodies Detect Survivin Cell Surface Expression and Inhibit Tumor Growth In Vivo. Clin Cancer Res. 2018 Jun 1;24(11):2642-2652. doi: 10.1158/1078-0432.CCR-17-2778. Epub 2018 Mar 14. PMID 29540489
- [Result] Rohayem J, Diestelkoetter P, Weigle B, Oehmichen A, Schmitz M, Mehlhorn J, Conrad K, Rieber EP. Antibody response to the tumor-associated inhibitor of apoptosis protein survivin in cancer patients. Cancer Res. 2000 Apr 1;60(7):1815-7. PMID 10766164
- [Result] Fenstermaker RA, Ciesielski MJ, Qiu J, Yang N, Frank CL, Lee KP, Mechtler LR, Belal A, Ahluwalia MS, Hutson AD. Clinical study of a survivin long peptide vaccine (SurVaxM) in patients with recurrent malignant glioma. Cancer Immunol Immunother. 2016 Nov;65(11):1339-1352. doi: 10.1007/s00262-016-1890-x. Epub 2016 Aug 30. PMID 27576783
- [Result] Adida C, Crotty PL, McGrath J, Berrebi D, Diebold J, Altieri DC. Developmentally regulated expression of the novel cancer anti-apoptosis gene survivin in human and mouse differentiation. Am J Pathol. 1998 Jan;152(1):43-9. PMID 9422522
- [Result] Sasaki T, Lopes MB, Hankins GR, Helm GA. Expression of survivin, an inhibitor of apoptosis protein, in tumors of the nervous system. Acta Neuropathol. 2002 Jul;104(1):105-9. doi: 10.1007/s00401-002-0532-x. Epub 2002 Mar 29. PMID 12070671
- [Result] Fukuda S, Pelus LM. Survivin, a cancer target with an emerging role in normal adult tissues. Mol Cancer Ther. 2006 May;5(5):1087-98. doi: 10.1158/1535-7163.MCT-05-0375. PMID 16731740
- [Result] Zaffaroni N, Daidone MG. Survivin expression and resistance to anticancer treatments: perspectives for new therapeutic interventions. Drug Resist Updat. 2002 Apr;5(2):65-72. doi: 10.1016/s1368-7646(02)00049-3. PMID 12135582
- [Result] Luoto S, Hermelo I, Vuorinen EM, Hannus P, Kesseli J, Nykter M, Granberg KJ. Computational Characterization of Suppressive Immune Microenvironments in Glioblastoma. Cancer Res. 2018 Oct 1;78(19):5574-5585. doi: 10.1158/0008-5472.CAN-17-3714. Epub 2018 Jun 19. PMID 29921698
- [Result] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT05163080/Prot_SAP_000.pdf